CLINICAL TRIAL: NCT04362007
Title: A Phase I/II, Multicenter, Open-Label, Nonrandomized Study to Evaluate the Tolerability and Safety of ASTX660 and the Efficacy at the Recommended Dose of ASTX660 in Patients With Relapsed or Refractory T-Cell Lymphoma
Brief Title: A Phase I/II Study of ASTX660 in Patients With Relapsed or Refractory T-cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to Sponsor decision, the decision to terminate was not based on any safety concerns.
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 401-102-00001; JapicCTI-205258 (Other Grant/Funding Number: Japic)
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-04

CONDITIONS: Relapsed or Refractory Peripheral T-cell Lymphoma(PTCL),Cutaneous T-cell Lymphoma(CTCL),Adult T-cell Leukemia/Lymphoma(ATLL)
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — ASTX-660

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 dose-escalation part (Experimental): Subjects with r/r PTCL and r/r CTCL will receive ASTX660 once a day for 7 consecutive days every other week of each 28-day cycle (ie, [7 days on/ 7 days off] ×2; daily dosing on Days 1-7 and 15-21). The starting dose will be escalated stepwise in successive cohorts of 3 to 6 evaluable subjects each (standard 3+3 study design), until the RD is determined.
  Interventions: Drug: ASTX660
- Phase 1 ATLL expansion part (Experimental): Subjects with r/r ATLL will receive ASTX660 at RD obtained from the Phase 1 part (dose-escalation part) once a day for 7 consecutive days every other week of each 28-day cycle.
  Interventions: Drug: ASTX660
- Phase 2 (Experimental): Subjects with r/r PTCL will receive ASTX660 at RD obtained from the Phase 1 part (dose-escalation part) once a day for 7 consecutive days every other week of each 28-day cycle.
  Interventions: Drug: ASTX660

INTERVENTIONS:
Drug: ASTX660 — Treatment of ASTX660 for r/r PTCL and r/r CTCL
  Arms: Phase 1 dose-escalation part
Drug: ASTX660 — Treatment of ASTX660 for r/r ATLL
  Arms: Phase 1 ATLL expansion part
Drug: ASTX660 — Treatment of ASTX660 for r/r PTCL
  Arms: Phase 2

SUMMARY:
Phase 1 (dose-escalation part): Investigate the tolerability and safety of ASTX660 in patients with r/r PTCL and r/r CTCL and determine the recommended dose (RD) for the Phase 2.

Phase 1 (ATLL expansion part): Evaluate the safety of ASTX660 at RD in patients with r/r ATLL.

Phase 2 : Evaluate the efficacy of ASTX660 at RD in patients with r/r PTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T-cell lymphoma with histological diagnosis based on WHO classification (2017)
2. Patients with evaluable lesions.
3. Patients with ECOG PS score of 0 or 1.
4. Patients with adequate organ functions as shown below.

   * AST and ALT ≤ 2.0 × ULN (≤ 3.0 × ULN if liver infiltration is present)
   * Total bilirubin ≤ 1.5 × ULN
   * ANC ≥ 1,000/mm3 (≥ 750/mm3 if bone marrow infiltration is present)
   * Platelet count 50,000/mm3 (25,000/mm3 if bone marrow infiltration is present)
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min
   * Amylase and lipase ≤ 1.0 × ULN

Exclusion Criteria:

1. Patients with active infection requiring treatment with antibiotics, antifungals, or antivirals
2. Patients with heart disease that meets the followings:

   1. LVEF of < 50% by echocardiography or MUGA scan
   2. Congestive heart failure (NYHA classification III or IV)
   3. Uncontrolled heart disease including unstable angina pectoris or hypertension considered to require hospitalization within last 3 months (90 days)
   4. Complete left bundle branch block, III degree (complete) atrioventricular block, use of pacemaker, history or complication of poorly controlled arrhythmia requiring treatment
   5. History or complication of long QT syndrome
   6. History or complication of ventricular arrhythmia requiring active treatment
   7. Corrected QT interval of ≥ 470 msec based on 12-lead ECG performed at the screening
   8. Concern on increased cardiac risk by participating in the study based on medical judgment
3. Patients receiving the following treatment for the primary disease prior to the initial dose of study drug

   1. Chemotherapy or radiotherapy within last 3 weeks
   2. Skin directed therapy including local treatment or phototherapy within last 3 weeks
   3. Treatment with monoclonal antibody within last 4 weeks
   4. Treatment with other study drugs or study treatment within last 3 weeks or 5 half-lives, whichever is longer
4. Patients with prior allogeneic stem cell transplantation, or autologous stem cell transplantation within 14 weeks prior to the day of initial dose of study drug
5. Patients who have received corticosteroids at a dose exceeding a prednisone equivalent dose of 10 mg/day within 3 weeks prior to the initial dose of study drug.
6. Patients with Inadequately controlled diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Safety (Phase 1 dose-escalation part) - number of subjects with dose-limiting toxicities (DLTs), AEs, abnormal clinical laboratory values or physical exam results | Up to 52.6 months
  Incidence of DLTs and other adverse events (AEs)
Safety (Phase 1 ATLL expansion part) - number of subjects with AEs, abnormal clinical laboratory values or physical exam results | Up to 52.6 months
  Incidence of adverse events (AEs)
Efficacy (Phase 2) - antitumor activity assessed by objective response rate (ORR) | Up to 52.6 months
  Antitumor activity by ORR by the Central Data Review Committee based on Lugano response criteria for non-Hodgkin's lymphoma by International Working Group (2014)

SECONDARY OUTCOMES:
Pharmacokinetic outcome of concentration-time curve (AUC) | Up to Day 1 in Cycle 2 (28 days per cycle)
  Assessment of pharmacokinetic parameter area under the concentration-time curve (AUC).
Pharmacokinetic outcome of maximum concentration (Cmax) | Up to Day 1 in Cycle 2 (28 days per cycle)
  Assessment of pharmacokinetic parameter maximum concentration (Cmax).
Pharmacokinetic outcome of time to maximum concentration (Tmax) | Up to Day 1 in Cycle 2 (28 days per cycle)
  Assessment of pharmacokinetic parameter time to maximum concentration (Tmax).
Pharmacokinetic outcome of samples over time | Up to Day 1 in Cycle 2 (28 days per cycle)
  Assessment of pharmacokinetic parameter elimination half life (t½).
Pharmacokinetic outcome of clearance of drug from plasma | Up to Day 1 in Cycle 2 (28 days per cycle)
  Assessment of pharmacokinetic parameter clearance of drug from plasma.
Common in all parts: antitumor activity assessed by ORR | Up to 52.6 months
  Antitumor activity by Investigator- or subinvestigator-assessed ORR
Common in all parts: antitumor activity assessed by duration of response (DOR) | Up to 52.6 months
  Time from the date of the earliest assessment of complete response or partial response to the date of relapse or death, whichever occurs earlier, or the last efficacy assessment date for subjects without a relapse or death.
Common in all parts: antitumor activity assessed by progression free survival (PFS) | Up to 52.6 months
  Number of days from the start of the study treatment to disease progression or death, whichever occurs first.
Common in all parts: overall survival (OS) | Up to 52.6 months
  Number of days from the day the subject received the first study treatment to the date of death, regardless of cause.
Common in all parts: time to response (TTR) | Up to 52.6 months
  Time from the day the subject received the first study treatment to the date of the earliest assessment of complete response or partial response.
Common in all parts: time to Progerssion (TTP) | Up to 52.6 months
  Time from the day the subject received the first study treatment to the date of relapse.
Common in all parts: Percentage of patients who switch to transplant | Up to 52.6 months
  Percentage of patients who switch to transplant
Safety (Phase 2) - number of subjects with AEs, abnormal clinical laboratory values or physical exam results. | Up to 52.6 months
  Incidence of adverse events (AEs)
Exploratory (Phase 1 dose-escalation part) - Assessment changes in cIAP in PBMC. | Up to 52.6 months
  Percentage degradation of cIAP1 protein in PBMCs from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Yamagata University Hospital, Yamagata, Japan

IPD SHARING:
Plan to Share IPD: No
The focus of this study is a rare disease.